CLINICAL TRIAL: NCT01666691
Title: Randomized, Double-Blind, Placebo Controlled, Dose Ranging Phase 2 Trial of Beloranib (ZGN-440 for Injectable Suspension), A Novel Methionine Aminopeptidase 2 Inhibitor, in Obese Subjects to Evaluate Weight Reduction, Safety, and Pharmacokinetics Over 12 Weeks
Brief Title: An Efficacy, Safety and Pharmacokinetics Study of Beloranib (ZGN-440 for Injectable Suspension) in Obese Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zafgen, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZAF-201
Record Dates: First submitted 2012-08-08; First posted 2012-08-16 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-07

CONDITIONS: Obesity
Keywords: Obese; Obesity; Overweight; Weight loss; Weight reduction; Beloranib
MeSH Terms: conditions — Obesity; Overweight; Weight Loss | interventions — CKD732

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Placebo (Placebo Comparator): ZGN-440 sterile diluent
  Interventions: Drug: Placebo
- 0.3 mg Beloranib (Experimental): 0.3 mg ZGN-440 for injectable suspension
  Interventions: Drug: Beloranib
- 0.6 mg Beloranib (Experimental): 0.6 mg ZGN-440 for injectable suspension
  Interventions: Drug: Beloranib
- 1.2 mg Beloranib (Experimental): 1.2 mg ZGN-440 for injectable suspension
  Interventions: Drug: Beloranib
- 2.4 mg Beloranib (Experimental): 2.4 mg ZGN-440 for injectable suspension
  Interventions: Drug: Beloranib
- 3.2 mg Beloranib (Experimental): 3.2 mg ZGN-440 for injectable suspension
  Interventions: Drug: Beloranib

INTERVENTIONS:
Drug: Beloranib — Subjects will receive ZGN-440 twice-weekly subcutaneous injections for up to 12 weeks and a total of 24 doses. A range of doses will be evaluated.
  Other Names: ZGN-440 for injectable suspension; ZGN-440; ZGN-433
  Arms: 0.3 mg Beloranib; 0.6 mg Beloranib; 1.2 mg Beloranib; 2.4 mg Beloranib; 3.2 mg Beloranib
Drug: Placebo — Subjects will receive placebo twice-weekly subcutaneous injections for up to 12 weeks and a total of 24 doses.
  Other Names: ZGN-440 sterile diluent
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate weight reduction, safety and pharmacokinetics for certain doses of beloranib (ZGN-440 for injectable suspension) administered as twice-weekly subcutaneous injections for 12 weeks.

DETAILED DESCRIPTION:
This protocol is designed to test the safety and efficacy of a drug called beloranib (ZGN-440 for injectable suspension). It is to be tested for its ability to reduce weight in obese subjects. The study will provide information on how much ZGN-440 gets into the blood, how long it stays in the body, and how it affects other biological markers.

ELIGIBILITY:
Inclusion Criteria:

* Obese volunteers weighing ≥ 50 kg
* BMI ≥ 30 and ≤ 50 kg/m2
* Stable body weight during the past 2 months
* Type 2 diabetes mellitus is allowed

Exclusion Criteria:

* Use of weight loss agents in the past month
* Current, clinically significant eating disorder
* Type 1 diabetes mellitus

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2012-08; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of beloranib (ZGN-440 for injectable suspension) administered subcutaneously for 12 weeks | Up to 26 weeks
  Safety and tolerability of beloranib will be assessed by comparing frequency and severity of adverse events as well as changes in physical examinations, ECGs, vital signs and laboratory evaluations. Other safety oriented questionnaires and parameters (e.g. sleep quality, hemodynamic parameters) will be measured and evaluated.
Weight loss and responses in metabolic biomarkers over a dose range of ZGN-440 | Up to 13 weeks
  Change from baseline in body weight and body composition (bioimpedance assessments), and scores of hunger/appetite over the dosing period will be evaluated to document beloranib's effect on obesity. Biomarkers of lipid metabolism will be measured to assess possible mechanisms of loss of body fat, as well as endocrinologic or anti-inflammatory markers.

SECONDARY OUTCOMES:
Pharmacodynamics over a dose range of beloranib | Up to 12 weeks
  The plasma PK of beloranib and selected metabolites may be assessed following dose administration to compare systemic exposure and PK parameters over the range of doses. PK parameters include Cmax, Tmax, AUC24hour, AUC∞, volume of distribution, total clearance, terminal elimination constant, and half-life. Mean residence time may also be reported.
Compare the plasma pharmacokinetic profile of beloranib administered subcutaneously with the profiles obtained previously using an alternative formulation administered subcutaneously and with ZGN-433 (beloranib hemioxalate) administered intravenously | Up to 12 weeks
Apparent bioavailability over a dose range of beloranib | Up to 12 weeks
  Bioavailability will be estimated from the SC PK parameters compared to the profile from comparable doses in earlier IV administration studies.

CONTACTS AND LOCATIONS:
Overall Officials: J K Marjason, MD, Principal Investigator — Q-Pharm Clinics, Royal Brisbane and Women's Hospital
Locations (3):
- Australia (3):
  - Q-Pharm Clinics, Royal Brisbane and Women's Hospital, Brisbane, Queensland
  - CMAX, Adelaide, South Australia
  - Linear Clinical Research Ltd, Perth, Western Australia